CLINICAL TRIAL: NCT00324519
Title: Randomized Trial Comparing Misoprostol and Foley Bulb for Pregnancy Termination in the Second Trimester
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-2005
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Pregnancy Trimester, Second; Induced Abortion
Keywords: second trimester; pregnancy termination; misoprostol; foley bulb
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Misoprostol Drug (Active Comparator): This is the misoprostol drug.
  Interventions: Drug: misoprostol
- The Foley Bulb (Experimental): This is the experimental portion to test the Foley Bulb.
  Interventions: Device: Foley bulb

INTERVENTIONS:
Device: Foley bulb
  Arms: The Foley Bulb
Drug: misoprostol
  Arms: Misoprostol Drug

SUMMARY:
The purpose of this study is to compare two methods of pregnancy termination on the time to delivery in the second trimester.

DETAILED DESCRIPTION:
Medical termination in the second trimester is performed for many indications. Successful termination is dependant on ripening of the cervix prior to labor induction. Multiple methods of cervical ripening and labor induction have been used for pregnancy termination in the second trimester. These two methods have different mechanisms of action. This study seeks to evaluate the effectiveness of these two methods.

ELIGIBILITY:
Inclusion Criteria:

* indication for pregnancy termination, gestational age from 13-27 weeks

Exclusion Criteria:

* multiple gestation, previous uterine surgery, rupture of membranes, latex allergy

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2005-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Time to vaginal delivery

SECONDARY OUTCOMES:
Rate of chorioamnionitis
Rate of maternal fever
Rate of postpartum hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Keri A Baacke, MD, Principal Investigator — University of Florida
Locations (1):
- Shands Hospital at the University of Florida, Gainesville, Florida, United States